CLINICAL TRIAL: NCT05103423
Title: A Multicenter, Randomized, Double-blind, Placebo Parallel-controlled, Phase I/II Study to Explore Safety and Efficacy of BDB-001 Injection in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Safety and Efficacy Study of BDB-001 Injection in Patients With Moderate to Severe Hidradenitis Suppurativa (HS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STS-BDB001-06
Record Dates: First submitted 2021-06-23; First posted 2021-11-02 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-06

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — BDB001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group 1 (Experimental)
  Interventions: Drug: BDB-001 Injection; Drug: Placebo
- Treatment group 2 (Experimental)
  Interventions: Drug: BDB-001 Injection; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BDB-001 Injection — Multiple IV infusions of BDB-001 Injection diluted in sodium chloride
  Arms: Treatment group 1; Treatment group 2
Drug: Placebo — Multiple IV infusions of Placebo Injection diluted in sodium chloride
  Arms: Treatment group 1; Treatment group 2
Drug: Placebo — Multiple IV infusions of Placebo Injection diluted in sodium chloride
  Arms: Placebo

SUMMARY:
A study to explore the safety and efficacy of treatment with BDB-001 Injection in adults with moderate to severe hidradenitis suppurativa (HS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old≤Age≤65 years old, male or female;
* Diagnosis of HS for at least 6 months;
* HS lesions must be present in at least two distinct anatomical areas, one of which must be at least located in the apocrine sweat gland area and Hurley Stage II or Hurley Stage III;
* Total abscess and inflammatory nodule (AN) count of ≥ 3.

Exclusion Criteria:

* Subject was previously treated with adalimumab or another biologic product during the 3 months before the first administration;
* Subject received any oral antibiotic treatment for HS within 2 weeks before the first administration;
* Subject received any oral retinoids treatment for HS within 4 weeks before the first administration;
* Subject received oral opioids analgesics within 1 week before the first administration;
* Systematic treatment with glucocorticoid or intramural injection within 4 weeks before the first administration;
* History of heart disease or malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | Week 8
  Safety and tolerability of BDB-001 injection after multiple administration in the treatment of HS patients.
Number of Participants developing anti-BDB-001 antibodies. | Week 8
  Safety and tolerability of BDB-001 injection after multiple administration in the treatment of HS patients.
Area under the plasma concentration versus time curve (AUC) of BDB-001 Assessment of pharmacokinetic parameters. | Week 8
  To evaluate the pharmacokinetic characteristics of BDB-001 injection after multiple administration in HS patients.
Peak Plasma Concentration (Cmax) of BDB-001and time to reach Cmax Assessment of pharmacokinetic parameters. | Week 8
  To evaluate the pharmacokinetic characteristics of BDB-001 injection after multiple administration in HS patients.
Minimal Plasma Concentration (Cmin) of BDB-001 Assessment of pharmacokinetic parameters. | Week 8
  To evaluate the pharmacokinetic characteristics of BDB-001 injection after multiple administration in HS patients.
Terminal phase half-life Assessment of pharmacokinetic parameters. | Week 8
  To evaluate the pharmacokinetic characteristics of BDB-001 injection after multiple administration in HS patients.

SECONDARY OUTCOMES:
Change in International Hidradenitis Suppurativa Severity Score System (IHS4) score from Day 0 by time point | From Day 0 until Day 56
  The International Hidradenitis Suppurativa Severity Score 4 (IHS4: developed by the European Hidradenitis Suppurativa Foundation Investigator Group)，IHS4 Score=(Nodule Count) + (Abscess Count*2) + (Draining Tunnel Count *4).
  IHS4 score uses a range grades:
  Mild= 0-3; Moderate=4-10; Severe ≥11.
Change in modified Sartorius Score (mSS) from Day 0 by time point | From Day 0 until Day 56
  The mSS is a summation of HS lesions based on a number of factors including anatomical region, number and type of lesions, distance between relevant lesions and lesions clearly separated by normal skin in each region measured as HS clinical parameters. The scale title for mSS is points. The mSS has a minimum value of 0 and no upper limit. The higher the score the more severe is the disease/worse is the outcome.
Change in Hidradenitis Suppurativa Clinical Response (HiSCR) from Day 0 by time point | From Day 0 until Day 56
  The definition for response to treatment based on HiSCR relative to Baseline was: at least 50% reduction in abscesses and inflammatory nodule (AN) count (over all anatomical regions) with no increase in number of abscesses and in number of draining fistulas.
Change in Hidradenitis suppurativa-Physician Global Assessment (HS-PGA) score from Day 0 by time point | From Day 0 until Day 56
  Hidradenitis Suppurativa - Physician's Global Assessment (HS-PGA)classifies patients' severity into six categories:clear, minimal, mild, moderate, severe, and very severe, based on the number and quality of inflammatory lesions.
Changes of active lesions (number of inflammatory nodules, abscesses, fistulas, and abscess overflow score) from Day 0 by time point | From Day 0 until Day 56
Change in Dermatology Life Quality Index (DLQI) score from Day 0 by time point | From Day 0 until Day 56
  A score is documented for each of the 10 DLQI items, ranging from 0 to 3 for each item. The scale title for DLQI is points. The total score is the sum of the responses to all 10 DLQI items, ranging from the minimum of 0 points to the maximum of 30 points. A higher score corresponds to worse health related quality of life/outcome.
Changes in Pain VAS score from Day 0 by time point | From Day 0 until Day 56
  Pain VAS:This is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10) that best reflects the intensity of their pain. The scale title for the VAS is points. The minimum score is 0 points (No skin pain), and the maximum score is 10 points (Skin pain as bad as you can imagine). The higher the score the more severe is the disease/worse is the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Baoxi Wang, Master, Principal Investigator — Plastic Surgery Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (15):
- China (15):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Plastic Surgery Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Chinese Academy of Medical Sciences and Peking Union Medical College, Nanjing, Jiangsu
  - The First Hospital of Jilin Universitv, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No